CLINICAL TRIAL: NCT05670964
Title: EValuation of the Impact of the UPLUG DEvice Onto the iNfection Rate of Indwelling Central Venous Catheters in Patients Undergoing Chronic hEmodialysis
Acronym: UPLUG-EVIDENCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: liquidation of the compagny
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP211510
Record Dates: First submitted 2022-12-09; First posted 2023-01-04 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Renal Disease, Chronic; Hemodialysis Catheter Infection
Keywords: Central venous catheter; UPLUG; Infection
MeSH Terms: conditions — Renal Insufficiency, Chronic; Infections

STUDY DESIGN:
Intervention Model Description: Multi-centered open labelled two-arm randomized (1:1) superiority trial. One arm will have standard dialysis, the other arm will have dialysis using the UPLUG device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UPLUG Arm (Experimental): Patients will have regular central veinous catheter and UPLUG device for their dialysis sessions.
  Interventions: Device: Connecting valve system; Device: Central haemodialysis Venous Catheter
- Standard Of Care Arm (Other): Patients will have regular central veinous catheter (standard of care) for their dialysis.
  Interventions: Device: Central haemodialysis Venous Catheter

INTERVENTIONS:
Device: Connecting valve system — UPLUG Port (changed every 29 days) and UPLUG Disposable (changed at every dialysis session) ensure the connection between a regular haemodialysis catheter and an extracorporeal circuit, and proceed to different steps of haemodialysis session without handling the Luer-Lock connectors of the haemodialysis catheter
  Other Names: UPLUG Port; UPLUG Disposable
  Arms: UPLUG Arm
Device: Central haemodialysis Venous Catheter — Central haemodialysis venous catheter (CE marked) will be used within the scope of their intended purpose during the dialysis session

SUMMARY:
Infections are common complications among patients on chronic haemodialysis. Haemodialysis patients with a catheter have a 2- to 3-fold increased risk of hospitalization for infection and death compared with patients with an arteriovenous fistula or graft [0].

As it is a major concern for the medical community, this clinical investigation aims at assessing, in real world conditions, the impact of the UPLUG device onto the infection rate of indwelling central venous haemodialysis catheters.

UPLUG-EVIDENCE is an international, multicenter, randomised, open label trial that will evaluate the efficacy of the UPLUG device on the reduction of bacterial infections in patients undergoing chronic haemodialysis with central venous catheter (CVC).

The UPLUG device has been designed to :

1. reduce the haemodialysis catheter openings, hence potentially reducing the infectious risk,
2. improve the lock solution infusion using a positive pressure, limiting the thrombosis risk and associated haemodialysis catheter dysfunction
3. limit the time needed to connect and disconnect the patient, by facilitating how the different steps are operated, and even allowing a connection/disconnection with a single healthcare professional
4. ultimately enhance patient's autonomy with ergonomics & safe procedures

DETAILED DESCRIPTION:
A total of 464 end stage renal disease patients undergoing chronic haemodialysis and receiving a new (de novo or replacement) indwelling CVC will be randomly assigned in a 1:1 ratio to perform either standard-of-care dialysis (232) or standard-of-care dialysis associated with the UPLUG device (232).

The UPLUG device consists of 2 parts :

1. the UPLUG Port, a sterile, single use device connected to the distal Luer-Lock connectors of a regular central venous catheter. It may be connected up to 29 days and
2. the UPLUG Disposable, a sterile, single use device indicated for use with the UPLUG Port to perform a chronic haemodialysis therapy. it will be changed at every dialysis session.

Treatment period (16 weeks):

W1:D1 : first connection of the UPLUG Port The patient will be seen by a nurse or an investigator at D29, D57 and D85 for UPLUG port periodical replacement, and at D113 for the definitive withdrawal of the UPLUG port.

Follow-up period (29 days):

A last visit (onsite or call) is planned during the definitive withdrawal of the CVC or no later than 29 days after the end of the treatment period (D113) to assess the safety and well-being of the patient

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease
* Chronic haemodialysis
* indwelling de novo or replacement central veinous catheter

Exclusion Criteria:

* Life expectancy < 1 year
* Renal transplantation already scheduled at inclusion (living donor)
* Current infection of CVC percutaneous or subcutaneous site
* Pregnant or breastfeeding female, or women without a medically significant contraceptive regimen
* Patient with mechanical heart valve
* Patient with an AVF likely to be functional within 1 month
* Strictly more than 3 dialysis sessions a week
* Patient undergoing haemodialysis session > 4h30
* Participation to another clinical study in the last 30 days period
* Patient unable to give a freely-given, written, informed consent
* Vulnerable participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Number of bacterial infection within the 16 weeks of treatment period | 16 weeks
  A clinical suspicion of bacterial infection is defined by :
  1/ fever (T>37.5°C) or Or 2/ rigor Or 3/ new pre-HD hypotension (systolic arterial pressure <90mmHg) Or 4/ confusion and/or disorientation at the investigator's discretion
  and will lead to a confirmation of bacteraemia**:
  Blood culture (BC) growing the same organism from :
  1/ HD catheter and 2a/ Peripheral vein And/or 2b/ Dialysis bloodline

SECONDARY OUTCOMES:
Number of clinical suspicion of bacterial infection during the 16 weeks of the treatment period, evaluated at Day 29, Day 57, Day 85 and Day 113 | Day 29, Day 57, Day 85 and Day 113
  A clinical suspicion of bacterial infection is defined by one of the following :
  1/ fever (T>37.5°C) Or 2/ rigor Or 3/ new pre-HD hypotension (systolic arterial pressure <90mmHg) Or 4/ confusion and/or disorientation at the investigator's discretion
Number of positive blood culture during the 16 weeks of the treatment period evaluated at Day 29, Day 57, Day 85 and Day 113 | Day 29, Day 57, Day 85 and Day 113
  Positive blood culture from one of the following :
  1/ HD catheter Or 2/ Peripheral vein Or 3/ Dialysis bloodline
Number of dysfunction estimated by blood flow rate (Qb) evaluated at Day 29, Day 57, Day 85 and Day 113 | Day 29, Day 57, Day 85 and Day 113
  Dysfunction is defined as:
  Qb < 200 ml/min during 30 minutes in the course of one haemodialysis session; Or Mean Qb < 250 ml/min during two consecutive haemodialysis sessions"
Number of adverse events during the 16 weeks of treatment period evaluated at D29, D57, D85 and D113 | D29, D57, D85 and D113
  Adverse events defined as defectiveness of the device, defectiveness of the placement, thrombosis events and infections
Number of infections other than bacterial during the 16 weeks of treatment period evaluated at Day 29, Day 57, Day 85 and Day 113 | Day 29, Day 57, Day 85, Day 113
  Infections other than bacterial : viral, fungal, parasitic
The patient satisfaction | Day 1, Day 29, Day 57, Day 85, Day 113, Day 141
  Patient satisfaction is assessed through :
  a specific UBIPLUG questionnaire and a questionnaire SF-36 (Short-Form 36 Health Survey)
Number of patients with at least one bacterial infection during the 16 weeks of treatment period evaluated at Day 29, Day 57, Day 85 and Day 113 | Day 29, Day 57, Day 85, Day 113
  A clinical suspicion of bacterial infection is defined by :
  1/ fever (T>37.5°C) or Or 2/ rigor Or 3/ new pre-HD hypotension (systolic arterial pressure <90mmHg) Or 4/ confusion and/or disorientation at the investigator's discretion
  and will lead to a confirmation of bacteraemia:
  Blood culture (BC) growing the same organism from :
  1/ HD catheter and 2a/ Peripheral vein And/or 2b/ Dialysis bloodline
Rate of infections other than bacterial evaluated at Day 29, Day 57, Day 85 and Day 113 | Day 29, Day 57, Day 85, Day 113
  infections other than bacterial : viral, fungal, parasitic
Rate of unplanned hospitalisation at Day 113 and at the end of the study | Day 113, Day 141
  Unplanned hospitalisation including less than 12 hours
Time spent by session by the nurse to connect the patient at Day 1, Day 29, Day 57, Day 85 and Day 113 | Day 1, Day 29, Day 57, Day 85, Day 113
  Measured time from the start of the catheter management to the start of the dialysis session
The nurse satisfaction for the patients in UPLUG arm | Day 1, Day 113
  Assessed through a specific UBIPLUG questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Hafedh FESSI, PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Dominique JOLY, PUPH, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Tenon, service de Néphrologie, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided